CLINICAL TRIAL: NCT04780282
Title: Effect of Scapular Stabilization Exercises on Proprioception, Muscle Strength, Disability and Throwing Performance in Water Polo Players
Brief Title: Effects of Scapular Stabilization Exercises on Water Polo Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ceren Çetin, Principal Investigator, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1614823
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Sport Injury
Keywords: exercise; muscle strength; physical performance; proprioception; sports injury
MeSH Terms: conditions — Motor Activity; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: It will be divided into 2 groups as scapular stabilization exercise group and control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular Stabilization Group (Experimental): In the study, Adalar Water Sports Club (AWSK) takes places with its A team players; 15 players aged from 16-25 as the scapular stabilization group. The players in the scapular stabilization group will be applied scapular stabilization exercises for 8 weeks, 3 days a week in company with a physiotherapist. As stabilization exercises for the players; 1)Squatting while sliding a towel on the wall, 2)Wall push-ups with one leg extension, 3)Cross squat, 4)Pulling elastic band while squatting on one leg, 5)Double-leg squatting
  Interventions: Other: Scapular Stabilization Group
- Control group (No Intervention): No Intevention

INTERVENTIONS:
Other: Scapular Stabilization Group — Participants will apply the 5 exercises given.
  Arms: Scapular Stabilization Group

SUMMARY:
30 water polo players will be included in this study. It will be divided into 2 groups as the scapular stabilization exercise group and the control group. Scapular stabilization exercise group;

1) Squat with a towel slide on the wall 2) Wall push-ups with one leg extension 3) Cross squat 4) Elastic band pull while one leg squats 5) Double leg squat exercises will be given. These exercises will be 8 weeks and 3 days a week. The measurements of the exercises will be taken before the first session and at the end of the last session of the 8th week. Without giving exercise to the control group, only measurements will be taken in the 1st and 8th weeks. The study will take place in Burhan Felek Swimming Pool. Measurement evaluation tests;

1. Arm, Shoulder and Hand Problems Questionnaire (DASH): It is a questionnaire used to determine the levels of upper extremity functionality.
2. Proprioception measurement: Digital goniometer device, which includes the use of constant gravity as a reference point to evaluate joint mobility, will be considered as active and passive repetitive positioning.
3. Measurement of muscle strength: The measurement will be made using a hand-held manual dynamometer J-TEC for isometric muscle strength evaluation.
4. Sitting medicine ball throwing (OSTA): The distance the participant throws the ball while in the long sitting position will be measured in "meters".

Statistical analysis to be used in the research will be done with SPSS 20.0 package program (SPSS inc, Chicago, USA).

DETAILED DESCRIPTION:
Water polo is a high-intensity team sport that originated in England in the 1860's as a sort of water rugby. The national team of water polo, which is one of the oldest team sports included in the Olympic programme, was formed in our country in 1934. Water polo is a sports branch in which basic and auxiliary biomotor skills are used high level in accordance with its technical and tactical features. Water polo players; are performing actions which consist of a combination of movements such as rising, diving, blocking, sprinting, controlling the ball, agility and shooting. The most important action among major movements that determines the result of the match is the skill of shooting. Water polo training, swimming, scissors, shooting and passing. After all of these, the players continue the technical-tactical team training in the water for the matches.

The essential physical suitability parameters of water polo players during performance are muscle endurance, flexibility,joint stabilization, muscular strength, muscle-strength balance and skills specific to water polo. It has been suggested that, in the case of weakness in these basic parameters, a risk factor for pain and injury may occur. The mostly injured parts of water polop players are; shoulder, hand, head, elbow and groin respectirely. It was reported that 13% of 260 water polo players were injured in London Summer Olympic Games(2012). Water polo players have their injuries mostly in the shoulder area and the reason is; the shoulder area carries 70% of the whole body weight while the legs carry 30%. Considering this ratio, it is seen that the risk of injury is inevitable. Among teh risk factors for shoulder injuries there take place insufficient shoulder stabilizaiton, hypermobility, repetitive throwing, rapid rotational movements for grasping and defensive movements.

In determining the rate and strength of shooting, shoulder joint stabilization is important. To optimize the function of the shoulder, scapula supports optimal muscle activation, increases the muscle strength and transfers the muscle strength and energy through the kinetic chain during shoulder movements, the dynamic movement of the scapula increases the stability of the glenohumeral joint. Scapular stabilization exercises are neuromuscular control exercises which support the posterior curvature and external rotation of the scapula and aims to develop the stabilization of the scapula and the shoulder and improve the motor control usually including visual, verbal and kinesthetic feedback. Studies done in the literature have shown that scapular stabilization exercises reduce the pain and disability in shoulder problems and increase the strength of the muscle in shoulder area.

Proprioception is an important part of shoulder stability and neuromuscular control. Disruption of the proprioceptive system leads to malfunctions in muscular activity and badly affected joint stabilization. The joint, whose stabilization and protective muscular activity is impaired, becomes vulnerable to external traumas. Deficiencies in the proprioceptive sense have been associated with a decrease in sporting performance. Also, repetitive throwing activities increase the risk of injury in the shoulder complex by causing a short-term weakening in shoulder muscle strength and proprioceptive functions. It has been claimed that greater sensory acvity contributes to the motor control of the joint through improved proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Being a players of Adalar Water Sports Club
* Being in the age rande of 16-25
* Agreeing to participate in the research voluntarily

Exclusion Criteria:

* Not being a player of Adalar Water Sports Club
* Having a history of fracture in the shoulder area
* Having received physiotherapy in the shoulder elbow and wrist 6 months ago

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male A team players will be taken
Enrollment: 30 (Estimated)
Dates: Start 2021-02-28 (Actual); Primary Completion 2022-08-08 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | Change between baseline and 8 weeks
  In the first part of the questionnaire, there are 20 questions on physical competence and in the following, of the questionnaire there are 10 questions on pain and a total of 30 questions evaluating the functional and environmental limitation as a outcome of it. In the second part of the questionnaire, there is a module consists of 4 questions for athletes-musicians who want high performance. There are 5 answer options in each item. The scores resulting from the answers given for all items of the questionnaire will be summed up and calculated. When the score gets higheri the degree of disability also gets higher.
Proprioception Measurement | Change between baseline and 8 weeks
  Digital goniometer device, which includes the use of constant gravity as a reference point to evaluate joint mobility, will be considered as active and passive repetitive positioning. researcher will initially bring the extremity to the target angle and wait there for a minimum of ten seconds for the patient to recall this position. Then the extremity will be placed in the starting position. The patient will be asked to actively bring his extremity back to the target angle or passively bring it to the previously determined angle. The deviation from the target angle (angular error) will be recorded.
Muscle Strength Measurement | Change between baseline and 8 weeks
  The measurement will be made using a hand-held manual dynamometer J-TEC for isometric muscle strength evaluation. Measurement will be applied to shoulder area flexion-extension, abduction-adduction, internal rotation-external rotation muscle groups
Throwing medicine ball in sitting position | Change between baseline and 8 weeks
  The distance the participant throws the ball while in the long sitting position will be measured in 'meters'.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla ATAŞ BALCI, Assist Prof, Study Director — Bahçeşehir University
Locations (1):
- Burhan Felek Swimming Club, Istanbul, Üsküdar, Turkey (Türkiye)